CLINICAL TRIAL: NCT01669512
Title: Safety and Immunogenicity of ChAd63 ME-TRAP / MVA ME-TRAP Heterologous Prime Boost Malaria Vaccination Adjuvanted With Matrix M™
Brief Title: Adjuvanting Viral Vectored Malaria Vaccines With Matrix M
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC048
Record Dates: First submitted 2012-08-14; First posted 2012-08-21 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Malaria; Matrix M
Keywords: Malaria vaccine; Matrix M
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control Regimen (Active Comparator): ChAd63 ME-TRAP 5 x 1010 vp on Day 0 and MVA ME-TRAP 2 x 108 pfu on Day 56 6 Volunteers
  Interventions: Biological: Control Regimen
- Low Dose Matrix M Regimen (Experimental): ChAd63 ME-TRAP 5 x 1010 vp mixed with Matrix M-1 25μg on Day 0 and MVA ME-TRAP 2 x 108 pfu mixed with Matrix M-1 25μg on Day 56 8 Volunteers
  Interventions: Biological: Low Dose Matrix M Regimen
- Standard Dose Matrix M Regimen (Experimental): ChAd63 ME-TRAP 5 x 1010 vp mixed with Matrix M-1 50μg on Day 0 and MVA ME-TRAP 2 x 108 pfu mixed with Matrix M-1 50μg on Day 56 8 Volunteers
  Interventions: Biological: Standard Dose Matrix M Regimen

INTERVENTIONS:
Biological: Control Regimen — ChAd63 ME-TRAP 5 x 1010 vp on Day 0 and MVA ME-TRAP 2 x 108 pfu on Day 56
  Arms: Control Regimen
Biological: Low Dose Matrix M Regimen — ChAd63 ME-TRAP 5 x 1010 vp mixed with Matrix M-1 25μg on Day 0 and MVA ME-TRAP 2 x 108 pfu mixed with Matrix M-1 25μg on Day 56
  Arms: Low Dose Matrix M Regimen
Biological: Standard Dose Matrix M Regimen — ChAd63 ME-TRAP 5 x 1010 vp mixed with Matrix M-1 50μg on Day 0 and MVA ME-TRAP 2 x 108 pfu mixed with Matrix M-1 50μg on Day 56
  Arms: Standard Dose Matrix M Regimen

SUMMARY:
ChAd63 METRAP and MVA METRAP are investigational vaccines for malaria which have been studied in clinical trials for 4 years, and 10 years, respectively. These vaccines are inactivated viruses which have been modified so that they cannot reproduce in humans. Genetic information has been added to make them express proteins of the malaria parasite so that they stimulate an immune response against malaria. This trial examines whether a compound called Matrix M™ can be used in efforts to improve on how well the vaccines work at preventing malaria.

Matrix M™ is a vaccine adjuvant, a compound used to improve the immune responses to vaccines. In this trial, Matrix M™ will be combined with each of the vaccines. The objectives are to assess the safety of the vaccines when combined with Matrix M™, and to determine what effect Matrix M™ has on the immune responses to the vaccines.

We will assess the safety of the vaccines (ChAd63 METRAP combined with Matrix M™; and MVA METRAP combined with Matrix M™) by administering them to healthy volunteers and monitoring them for 6 months in total. Eight volunteers will receive the vaccines with the low dose of Matrix M™, eight will receive the vaccines with the standard dose of Matrix M™, and six volunteers will receive the vaccines alone as a comparison group. We will also look at what effect Matrix M™ has on the immune responses to the vaccines, as measured from blood tests. Volunteers will have study visits to the Clinical Centre for Vaccinology and Tropical Medicine on the Churchill Hospital site, Oxford, where they will have vaccinations, have blood taken to monitor safety and measure immune responses to vaccination, and be monitored for symptoms/side effects from vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 18 to 50 years
* Able and willing (in the Investigator's opinion) to comply with all study requirements
* Willing to allow the investigators to discuss their medical history with their General Practitioner
* For female volunteers, willingness to practice continuous effective contraception during the study
* For male volunteers, must use barrier contraception for 3 months from the day of any administration of Matrix M™
* Agreement to refrain from blood donation during the course of the study and for 6 months after the end of their involvement in the study
* Written informed consent

Exclusion Criteria:

* Participation in another research study involving an investigational product in the 30 days preceding enrolment, or planned use during the study period
* Prior receipt of an investigational malaria vaccine or any other investigational vaccine likely to impact on interpretation of the trial data
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections; and chronic (more than 14 days) immunosuppressant medication use within the past 6 months (inhaled and topical steroids are allowed)
* Pregnancy, lactation, or intention to become pregnant during the study
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine, e.g. egg products, Kathon
* History of clinically significant contact dermatitis Any history of anaphylaxis or hypersensitivity in relation to vaccination
* History or evidence of pre-existing autoimmune or antibody-mediated disease or laboratory evidence of possible autoimmune disease, defined as a positive antinuclear antibody (ANA) result at screening.
* Any history of malaria
* Travel to a malaria endemic region during the study period or within the six months preceding enrolment in the study with significant risk of malaria infection
* History of serious psychiatric condition that may affect participation in the study
* Any other serious chronic illness requiring hospital specialist supervision
* Suspected or known current alcohol abuse as defined by an alcohol intake of greater than 42 units every week
* Suspected or known injecting drug abuse in the five years preceding enrolment
* Seropositive for hepatitis B surface antigen (HBsAg)
* Seropositive for hepatitis C virus (antibodies to HCV)
* Any relevant history of cancer (excludes basal cell carcinoma of the skin and cervical carcinoma in situ)
* Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
* Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of study data

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2012-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
To assess the safety of ChAd63 ME-TRAP / MVA ME-TRAP heterologous prime boost vaccination adjuvanted with Matrix M™ | 24 weeks from first vaccination
  Analysis of all solicited and unsolicited local and general vaccine-linked adverse events (AEs) occurring in Low Dose Matrix M™ and Standard Dose Matrix M™ Group volunteers.

SECONDARY OUTCOMES:
Assess the effects of Matrix M™ on the immunogenicity of ChAd63 ME-TRAP / MVA ME-TRAP heterologous prime boost vaccination | 24 weeks from first vaccination
  Comparison of immunogenicity of the Matrix M™ - adjuvanted vaccination regimens, versus the Control regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hill, MD, Principal Investigator — University of Oxford
Locations (1):
- Centre for Clinical Vaccinology and Tropical Medicine, Oxford, Oxfordshire, United Kingdom

REFERENCES:
- [Derived] Venkatraman N, Anagnostou N, Bliss C, Bowyer G, Wright D, Lovgren-Bengtsson K, Roberts R, Poulton I, Lawrie A, Ewer K, V S Hill A. Safety and immunogenicity of heterologous prime-boost immunization with viral-vectored malaria vaccines adjuvanted with Matrix-M. Vaccine. 2017 Oct 27;35(45):6208-6217. doi: 10.1016/j.vaccine.2017.09.028. Epub 2017 Sep 21. PMID 28941620